CLINICAL TRIAL: NCT06101992
Title: Randomized Double-blind Controlled Clinical Trial: the Use of Mesoglycan vs Placebo in the Acute Phase of Hemorrhoidal Disease
Brief Title: Mesoglycan for Acute Hemorrhoidal Disease
Acronym: CHORMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Collaborators: Neopharmed Gentili S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SICCR23
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — mesoglycan

STUDY DESIGN:
Intervention Model Description: Randomized double-blind controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesoglycan (Active Comparator): According to randomization, patients will take mesoglycan mg 50 (heparan sulphate 47.5%, dermathan sulphate 35.5%, chondroitin sulfate 8.5%,slow heparin 8.5%, excipients: lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide, erythrosine) 4 capsules/day for 5 days and 2 capsules/day for 35 days
  Interventions: Drug: Mesoglycan
- Placebo (Placebo Comparator): According to randomization, patients will take placebo (lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate) 4 capsules/day for 5 days and 2 capsules/day for 35 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesoglycan — Mesoglycan capsules 50 mg are composed by heparan sulphate 47.5%, dermathan sulphate 35.5%, chondroitin sulfate 8.5%,slow heparin 8.5%, excipients: lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide, erythrosine
  Other Names: MES
  Arms: Mesoglycan
Other: Placebo — placebo capsules are composed by lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate
  Other Names: PLA
  Arms: Placebo

SUMMARY:
Hemorrhoidal disease (HD) is the most common proctological disease with a prevalence rate that can reach approximately 4.4% of the population, with a particular peak in individuals aged between 45 and 65 years. The most common presentation of HD is painless rectal bleeding occurring during or immediately after defecation. Pain is rare in case of uncomplicated HD and may be present in case of external hemorrhoidal thrombosis.

The decision-making to treat Hemorrhoidal thrombosis usually depends on the timing of the onset of symptoms, with the surgical treatment favored if the onset of symptoms occurs within 72 hours.

Mesoglycan, a natural preparation of glycosaminoglycans (GAGs), is a polysaccharide complex rich in sulfur radicals.

It is composed of heparan sulphate (47.5%), dermatan sulphate (35.5%), chondroitin sulfate (8.5%) and slow heparin (8.5%).

Mesoglycan exerts antithrombotic activity (activation of antithrombin III and heparin cofactor II) and profibrinolytic (stimulation of the activator tissue plasminogen) decreasing plasma concentrations of fibrinogen without affecting the prothrombin time, the time of partial thromboplastin or the remaining coagulation parameters. The rationale of this double-blind randomized controlled clinical trial is to confirm/evaluate the efficacy and safety of mesoglycan versus placebo in reducing the symptoms of hemorrhoidal disease and their impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade I-III hemorrhoidal disease classified according to Goligher classification or diagnosis of external hemorrhoid thrombosis
* Female patients of childbearing age with a negative pregnancy test
* Patients able to understand informed consent
* Signed Informed Consent.

Exclusion Criteria:

* Blood coagulations disorders
* Patients undergoing chemoradiation
* intake of anticoagulants
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms relief | 40 days
  According to the validated Hemorrhoidal Disease Symptom Score (from 0: no symptoms to 20: symptoms occurring every day), score reduction will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Arcangelo Picciariello, MD, Study Chair — Societa Italiana di Chirurgia ColoRettale

REFERENCES:
- [Derived] Gallo G, Picciariello A, Realis Luc A, Salvatore A, Di Vittori A, Rinaldi M, Trompetto M. Use of mesoglycan in the acute phase of hemorrhoidal disease (the CHORMES study): study protocol for a double-blind, randomized controlled trial. Trials. 2024 Dec 2;25(1):807. doi: 10.1186/s13063-024-08648-y. PMID 39623365